CLINICAL TRIAL: NCT02510651
Title: Effect of Procedural-Related Variables on Melanocyte-Keratinocyte Suspension Transplantation in Non-Segmental Stable Vitiligo: A Clinical and Immunohistochemical Study
Brief Title: Effect of Procedural Variables on Outcome of Surgical Treatment of Vitiligo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Abdel Halim, Assisstant professorof dermatology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAH555
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Vitiligo
Keywords: : non-segmental vitiligo; melanocyte-keratinocyte suspension; cryoblebbing; CO2 laser
MeSH Terms: conditions — Vitiligo | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ORSHFS (Experimental): Melanocyte-keratinocyte suspension.
  Interventions: Procedure: Melanocyte-keratinocyte suspension

INTERVENTIONS:
Procedure: Melanocyte-keratinocyte suspension — Treatment of non-segmental vitiligo by CO2 laser followed by melanocyte-keratinocyte suspension.
  Other Names: CO2 laser

SUMMARY:
ORSHFS grafts yielded lower cell counts than NCECS but the M-K ratio and resultant repigmentation did not show significant difference with better healing of the donor site. Compared to cryoblebs, CO2 gave more homogenous pigmentation. The acral sites showed better results using combination of donor NCECS and recipient cryoblebs.

DETAILED DESCRIPTION:
Background: Melanocyte-keratinocyte suspension (M-K susp) is gaining popularity for vitiligo treatment. Few studies have addressed procedure-related variables.

Objective: To assess the effect of different M-K susp procedure-related variables on the clinical outcome in stable vitiligo.

Methods: This retrospective study included 40 cases with stable non-segmental vitiligo treated by M-K susp followed by narrow band- ultraviolet B phototherapy twice weekly. Donor site was either a skin graft in non-cultured epidermal cell suspension (NCECS) (34 cases) or hair follicle unit in Outer Root Sheath Hair Follicle Suspension (ORSHFS) (6 cases). Recipient site was prepared by either cryoblebbing (24 cases) or carbon dioxide (CO2)laser resurfacing (16 cases). Cell counts and viability were recorded in the cell suspensions, and tissue melanocytes and keratinocytes were examined by Melan A and Cytokeratin respectively. Assessment of repigmentation was done 18 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Stable non-segmental vitiligo

Exclusion Criteria:

* Active vitiligo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The number of patients with satisfactory response after the surgical procedure for vitiligo. | one year